CLINICAL TRIAL: NCT05380843
Title: Description of Treatment Patterns and Population Characteristics of Pre-dialysis CKD Patients in the Czech Republic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Value Outcomes Ltd. (Other)
Responsible Party: Sponsor
Other Study IDs: NephroSCREEN
Record Dates: First submitted 2022-05-09; First posted 2022-05-19 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Chronic Kidney Diseases
Keywords: epidemiological survey; renal failure; decreased renal function; dialysis; low protein diet; treatment alternatives; Clinical Frailty Scale; Mini Nutritional Assessment (MNA); Bansal Score
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Insufficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The decision making in the Czech nephrology offices depends on the local common practice which is likely to be heterogenous. In other words, the same patient would be indicated to different therapy and regimen at different sites. To date, the practices and treatment paths have not been described. The aim of the present epidemiological research is to characterize the population of CKD patients at the point of treatment choice and to outline the motivation of nephrologist to initiate particular therapy.

DETAILED DESCRIPTION:
This is epidemiological (observational) cross-sectional survey. Data for the research will be obtained from clinical records and patient´s questionnaires and transcribed into electronic case report forms (eCRF) by physician anonymized using subject ID.

This observational research will not impose any additional procedures, assessments, or changes in addition to the routine management of subjects.

The research does not aim to follow treatment with a single medicinal product. The management of patients will be described in general terms. Names of active substances will be collected rather than the names of individual products.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient of 18 years and older
* Signed consent with processing of personal data as per the GDPR and the applicable national legal requirements
* Chronic kidney disease (CKD) category 4 to 5 characterized by GFR < 30 ml/min/1.73m2 for at least 3 months

Exclusion Criteria:

* Patients on chronic dialysis
* Patient waiting for kidney transplant
* Patient requiring indication of dialysis (e.g., life-threatening changes in fluid, electrolyte, and acid-base balance, serositis, pruritus, inability to control blood pressure, lethargy or other changes in mental status, symptoms of uraemia, GFR < 10 ml/min/1.73 m2)
* Patient with altered mental state unable to fill patient questionnaires

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with severely decreased renal function or with renal failure (CKD category 4 to 5 as per KDIGO 2012 (2), i.e., GFR < 30 ml/min/1.73 m2 for at least 3 months) naïve to dialysis.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Sociodemographic parameters | through study completion, an average of 3 months
  age, gender, ethnicity, health insurance company, education, marital status and cohabitation, employment status/disability, type of employment

SECONDARY OUTCOMES:
Medical history and anthropometry | through study completion, an average of 3 months
  BMI (in kg/m^2)
Medical history and anthropometry | through study completion, an average of 3 months
  blood pressure (systolic/diastolic, in mmHg)
Medical history and anthropometry | through study completion, an average of 3 months
  time since CKD diagnosis (in years), time since stage 4 CKD (in years), previous referral to nephrology (in years)
Medical history and anthropometry | through study completion, an average of 3 months
  smoking, abusus
Medical history and anthropometry | through study completion, an average of 3 months
  aetiology of CKD, comorbidities, current pharmacotherapy
Laboratory parameters | through study completion, an average of 3 months
  albumin (in g/l)
Laboratory parameters | through study completion, an average of 3 months
  glycaemia (in mmol/l)
Laboratory parameters | through study completion, an average of 3 months
  CRP (in mg/l)
Laboratory parameters | through study completion, an average of 3 months
  serum creatinine (in μmol/l)
Laboratory parameters | through study completion, an average of 3 months
  serum calcium (in mmol/l)
Laboratory parameters | through study completion, an average of 3 months
  LDL and HDL cholesterol (in mmol/l)
Laboratory parameters | through study completion, an average of 3 months
  serum urea (in mmol/l)
Laboratory parameters | through study completion, an average of 3 months
  plasma potassium (in mmol/l)
Laboratory parameters | through study completion, an average of 3 months
  serum PTH (pmol/l)
Laboratory parameters | through study completion, an average of 3 months
  albuminuria (in mg/l)
Laboratory parameters | through study completion, an average of 3 months
  serum phosphorus (mmol/l)
Laboratory parameters | through study completion, an average of 3 months
  haematuria (erythrocytes/μl)
Laboratory parameters | through study completion, an average of 3 months
  urine creatinine (mmol/l)
Laboratory parameters | through study completion, an average of 3 months
  blood count - WBC (10^9/l)
Laboratory parameters | through study completion, an average of 3 months
  blood count - RBC (10^12/l)
Laboratory parameters | through study completion, an average of 3 months
  blood count - MCV (fl)
Laboratory parameters | through study completion, an average of 3 months
  blood count - MCHC (g/l)
Laboratory parameters | through study completion, an average of 3 months
  blood count - HCT
Laboratory parameters | through study completion, an average of 3 months
  blood count - HGB (g/l)
Laboratory parameters | through study completion, an average of 3 months
  blood count - PLT (10^9/l)
Laboratory parameters | through study completion, an average of 3 months
  blood count - RDW (%)
Prognosis | through study completion, an average of 3 months
  Bansal score (min. 0, max. 17, higher score means the worse prognosis)
Functional status/frailty/performance | through study completion, an average of 3 months
  Clinical frailty scale (min. 1, max. 9, higher score means higher frailty)
Nutrition | through study completion, an average of 3 months
  nutritional status (Full MNA assessment), ketoanalogues, salt intake, protein intake, nutritional education (flyers, consultations etc.), attitude/future adherence to prescribed dietary restrictions
Decision of future management | through study completion, an average of 3 months
  Choice of future management (conservative management, conservative management with ketoanalogues, dialysis)
Physician attitude to the choice of therapy + reasons | through study completion, an average of 3 months
  Physician motivation/reasons for treatment choices
Patient attitude to the choice of therapy + reasons | through study completion, an average of 3 months
  Patient motivation/reasons for treatment choices

CONTACTS AND LOCATIONS:
Locations (5):
- Czechia (5):
  - FMC Nemocnice Mělník, Mělník, Central Bohemia
  - FMC Sokolov, Sokolov, Karlovarský kraj
  - Nemocnice Havlíčkův Brod, Havlíčkův Brod, Kraj Vysočina
  - Nemocnice Jihlava, Jihlava, Kraj Vysočina
  - Thetis Seirenia Brno, Brno, South Moravian

IPD SHARING:
Plan to Share IPD: No